CLINICAL TRIAL: NCT01126294
Title: Perioperative Analgesic and Anxiolytic Effect of Melatonin in Patients Undergoing Lumbar Laminectomy
Brief Title: Perioperative Melatonin in Lumbar Laminectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Dr. Philip Peng, University Health Network
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09-0172-B
Record Dates: First submitted 2010-05-17; First posted 2010-05-19 (Estimated); Last update posted 2010-05-19 (Estimated); Status verified 2010-04

CONDITIONS: Pain and Anxiety in Patients Undergoing Surgery for Lumbar Laminectomy.
Keywords: lumbar laminectomy, melatonin, perioperative, pain, anxiety, analgesia, VAS score
MeSH Terms: conditions — Pain; Anxiety Disorders; Agnosia | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Melatonin 5 mg (Experimental): Patients will receive 5 mg melatonin once the evening before surgery and then again at 90 minutes before surgery.
  Interventions: Dietary Supplement: 5 mg melatonin
- Melatonin 10 mg (Experimental): Patients will receive 10 mg melatonin once the evening before surgery and then again at 90 minutes before surgery.
  Interventions: Dietary Supplement: 10 mg melatonin
- Placebo (Placebo Comparator): Patients will receive placebo once the evening before surgery and then again at 90 minutes before surgery.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: 5 mg melatonin — Patients will receive 5 mg melatonin once the evening before surgery and then again at 90 minutes before surgery.
  Arms: Melatonin 5 mg
Dietary Supplement: 10 mg melatonin — Patients will receive 10 mg melatonin once the evening before surgery and then again at 90 minutes before surgery.
  Arms: Melatonin 10 mg
Dietary Supplement: Placebo — Patients will receive placebo once the evening before surgery and then again at 90 minutes before surgery.
  Arms: Placebo

SUMMARY:
Patients undergoing lumbar laminectomy surgery will receive either 5 or 10 mg melatonin or placebo once the evening before surgery and again 90 minutes before surgery. Pain and anxiety will be assessed over the 24 hour period following surgery.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 65 years old
* ASA status 1-3
* having lumbar laminectomy 2 to 3 levels with or without fusion

Exclusion Criteria:

* receiving emergent procedure
* surgery for neoplastic spine lesion
* allergy to melatonin or its non-medicinal ingredients
* allergy or contraindication
* BMI over 35 or or less than 20 kg/m2
* pregnancy or breastfeeding
* failure to provide informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-07 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Pain | 24 hours
  Pain will be assessed over a 24 hour period following surgery using a visual analogue scale
Anxiety | 24 hours
  Anxiety will be assessed over a 24 hour following surgery using visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: Philip Peng, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Madsen BK, Zetner D, Moller AM, Rosenberg J. Melatonin for preoperative and postoperative anxiety in adults. Cochrane Database Syst Rev. 2020 Dec 8;12(12):CD009861. doi: 10.1002/14651858.CD009861.pub3. PMID 33319916